CLINICAL TRIAL: NCT00100113
Title: Study of Interactions Between GBR 12909 and Cocaine
Brief Title: Assessment of Potential Interactions Between GBR 12909 and Cocaine - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CPU-0004-1
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-03

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — vanoxerine

INTERVENTIONS:
Drug: GBR 12909

SUMMARY:
The purpose of this study is to assess potential interactions between intravenous (IV) cocaine and 3 doses of GBR 12909.

DETAILED DESCRIPTION:
This is Phase 1, double-blind, placebo-controlled human laboratory clinical pharmacology study that will assess the potential interactions between IV cocaine and 3 escalating oral doses of GBR 12909. The primary objective is to determine safety of GBR 12909 administration and if there are significant interactions between GBR 12909 treatment concurrent with IV cocaine infusions.

ELIGIBILITY:
Inclusion Criteria:

* Must be within 20% ideal body weight and must weigh at least 45 kg.
* Must understand the study procedures and provide written informed consent.
* Must meet DSM-4 criteria and are non-treatment seeking at time of study.

Exclusion Criteria:

* Please contact study site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2004-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Cunningham, Ph.D., Principal Investigator — University of Texas Medical Branch - Galveston
Locations (1):
- U of Texas Medical Branch Galveston, Galveston, Texas, United States